CLINICAL TRIAL: NCT05251311
Title: A Mixed-Method Evaluation of the Impact of Social Risk Screening on Uptake of Social Assistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-018785
Record Dates: First submitted 2021-09-30; First posted 2022-02-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Low-income Populations; Social Determinants of Health

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Social worker that follows up with each participant will be blinded to randomization arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Risk Screening + Resource Map (Experimental): Participants randomized to the experimental arm will receive a social risk assessment tool followed by an electronic resource map
  Interventions: Behavioral: Social Risk Screening Tool; Other: Electronic Resource Map
- Resource Map (Active Comparator): Participants randomized to the active comparator group will receive only an electronic resource map
  Interventions: Other: Electronic Resource Map
- Resource Menu + Resource Map (Experimental): Participants randomized to this experimental arm will receive a social resource menu tool followed by an electronic resource map.
  Interventions: Behavioral: Resource Menu

INTERVENTIONS:
Behavioral: Social Risk Screening Tool — Investigators will use an adapted version of the evidence-based WE CARE screening tool, which assesses need in the 5 domains most frequently requested by our patient population: housing, transportation, child care, food security, and household heat and electricity. This tool was selected as it is evidence-based, takes fewer than 5 minutes to complete, is written at a 3rd grade reading level, and allows for differentiation between social risk and caregiver desire for assistance, as well as areas of "emergency" need.
  Arms: Social Risk Screening + Resource Map
Other: Electronic Resource Map — All participants will receive access to an electronic, geographically searchable resource map hosted on Aunt Bertha
  Arms: Resource Map; Social Risk Screening + Resource Map
Behavioral: Resource Menu — Participants randomized to this experimental arm will receive a social resource menu tool, which assess desire for social resources.
  Arms: Resource Menu + Resource Map

SUMMARY:
Children are disproportionately affected by the rise in poverty rates in the United States. Economic hardships can compromise child development, overall health, and the ability to succeed in school and in life. The current economic recession and racial disparities underscored by COVID19 have magnified this impact on children and hastened the already rapid growth of screening protocols for social risk factors- such as food and housing insecurity, financial strain, and unsafe environments-within pediatric health care. However, it remains unclear what effect standardized screening has on family perception of and engagement with resources. Current implementation momentum for screening protocols is outpacing research, and is raising concern among patient advocates for unintended harm-alienating families for fear of stigma or worse, and overpromising services that may not exist. Through a rigorous mixed-method approach, the proposed study will explore the impact of screening on acceptance, perception, and engagement with social resources among families with children. Furthermore, by leveraging the new technology of resource mapping as the method of resource referral, this study will provide insight regarding its effectiveness as a social needs assistance strategy. The knowledge gained will provide guidance for policymakers and other healthcare systems on how to integrate social risk interventions into healthcare delivery in order to maximize the benefit to children and families.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers presenting with a child to the pediatric clinical setting
* Child age 0-25

Exclusion Criteria:

* Engaged in complex care management services
* Child in critical condition
* Presenting to clinical setting specifically for social work intervention

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3949 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Resource Uptake By Search | 30 days
  total number of searches
Resource Uptake By Domain | 30 days
  number of searches by domain
Resource Engagement By Time | 30 days
  time spent on site
Resource Engagement By Saves | 30 days
  number of resources saved
Resource Engagement By Domain | 30 days
  number of resources saved by domain
Resource Utilization | 30 days
  rates of resource utilization
Resource Impact | 30 days
  perceived impact of resource use on social need measured by using a modified version of the WE CARE screening tool

SECONDARY OUTCOMES:
Perceived impact of screening on resource acceptance | up to 45 days
  Qualitative semi-structured interviews
Perceived impact of screening on resource perception | up to 45 days
  Qualitative semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Cullen, MD MPH MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown R, Cigarroa Kennedy S, Carranco Chavez E, Dumeng-Rodriguez J, Cullen D. Evaluation of a notes-based rapid qualitative analysis method to facilitate implementation. Implement Sci Commun. 2025 Mar 3;6(1):23. doi: 10.1186/s43058-025-00709-w. PMID 40033458